CLINICAL TRIAL: NCT06536556
Title: Effects of a Single Chemotherapy Administration on Skeletal Muscle of Breast Cancer Patients: Comparison of Paclitaxel vs Paclitaxel + Trastuzumab vs Paclitaxel + Carboplatine: the PROTECT-06 Bis Study
Acronym: PROTECT-06-bis
Status: Terminated | Type: Observational
Why Stopped: Recruitment sufficiant in term of statistical power
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-029
Record Dates: First submitted 2024-05-13; First posted 2024-08-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Protein turnover; Skeletal muscle deconditoning; Breast cancer; Chemotherapy; Muscle biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — muscle micro-biopsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TAX Group: Woman with early breast cancer receiving a first cycle of TAX
  Interventions: Other: First Assessment; Other: Second Assessment
- TAX+TRASTU Group: Woman with early breast cancer receiving a first cycle of TAX+TRASTU
  Interventions: Other: First Assessment; Other: Second Assessment
- TAX+CARBO Group: oman with early breast cancer receiving a first cycle of TAX+CARBO
  Interventions: Other: First Assessment; Other: Second Assessment

INTERVENTIONS:
Other: First Assessment — pre-treatment assessment
Other: Second Assessment — 4 days post-treatment assessment

SUMMARY:
This study aims to investigate the acute effects (i.e. 4 days) of paclitaxel or paclitaxel vs trastuzumab or paclitaxel and carboplatine on skeletal muscle of breast cancer patients. Muscle biopsies will be performed, as well as measurements of body composition strength, muscle architecture and quality of life.

DETAILED DESCRIPTION:
Breast cancer patients are commonly treated with chemotherapy, which is known to induce severe side effects such as skeletal muscle deconditioning, characterized by skeletal muscle atrophy and major mitochondrial alterations. These maladaptations, observed in patients treated with epirubicin-cyclophosphamide (EC) followed by weekly paclitaxel (TAX), ultimately lead to reduction in exercise capacity and quality of life. However, little is known about the specific effect of each type of chemotherapy.

In our recent article (see Citations field in the References module), The investigators demonstrated that chemotherapy effects on skeletal muscle are drug-dependent. Using muscle biopsies before and 4 days after the first administration of EC or TAX, we demonstrated that unlike TAX, EC induced severe muscle atrophy and mitochondrial alterations. Of note, patients in the TAX group had already received EC during the preceding weeks (Figure 1). Therefore, these patients had already begun to have altered skeletal muscle homeostasis, which might have limited the influence of TAX compared with that of its administration in isolation (i.e., without other previous chemotherapy administrations). In addition, some patients had received, concomitantly with TAX, Trastuzumab (TRASTU) due to HER tumor mutation. Also, in triple negative breast cancers, the recommendations concerning neo(adjuvant) chemotherapy have recently changed and recommend starting treatment with the use of paclitaxel + carboplatin (TAX + CARBO).

ELIGIBILITY:
Inclusion Criteria:

TAX group :

* Female ≥ 18 years
* Stage I to III breast cancer
* Patient who has not yet started treatment with TAX
* Enrolled in a social security scheme
* Able to speak, read and understand French

TAX+TRASTU group :

* Female ≥ 18 years of age
* Stage I to III breast cancer
* Patient who has not yet started treatment with TAX+TRASTU (Tolaney regimen)
* Enrolled in a social security scheme
* Able to speak, read and understand French

Exclusion Criteria:

* Prior exposure to chemotherapy
* Musculoskeletal disorders, autoimmune, vascular or neuromuscular disease
* Implantation of a pacemaker
* Contraindications to fitness evaluation
* Contraindication to local anesthesia for microbiopsy
* Minor or protected adult
* Pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early-stage breast cancer receiving chemotherapy. It is planned to include a first group of 10 patients receiving their first administration of TAX and a second group of 10 patients receiving their first administration of TAX+TRASTU. A first session of assessments will take place before the first TAX or TAX+TRASTU session, and a second session 4 days (D4) after the session.
  It is planned to include the same number of patients per group, i.e. 10 patients per group, for a total of 20 patients in the study
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
To investigate the effects of a chemotherapy session on mitochondrial function of skeletal muscle in breast cancer patients by comparing the first session of TAX to the first session of TAX + TRASTU or +CARBO. | Change at 4 days post-treatment compare to baseline
  difference of a score combining the mitochondrial respiratory capacity with production of hydrogen peroxide, difference in protein levels (western blots) and mRNA (RT-qPCR) expression.

SECONDARY OUTCOMES:
Compare the effect of the first TAX to the first TAX+TRASTU or +CARBO on muscle fiber cross-sectional area;cellular mechanisms of inflammation,fat infiltration and protein turnover;body composition;strength;muscle architecture and quality of life | Change at 4 days post-treatment compare to baseline
  difference of a score combining the mitochondrial respiratory capacity with production of hydrogen peroxide, difference in protein levels (western blots) and mRNA (RT-qPCR) expression.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de cancérologie Strasbourg europe, Strasbourg, France

REFERENCES:
- [Background] Mallard J, Hucteau E, Bender L, Charlot A, Debrut L, Pflumio C, Trensz P, Schott R, Favret F, Pivot X, Hureau TJ, Pagano AF. Development of skeletal muscle atrophy and intermuscular adipose tissue in patients with early breast cancer treated with chemotherapy. Am J Physiol Cell Physiol. 2022 Oct 1;323(4):C1325-C1332. doi: 10.1152/ajpcell.00373.2022. Epub 2022 Sep 12. PMID 36094434